CLINICAL TRIAL: NCT06866899
Title: Comparison of Axillary Block Regional Anesthesia and Wide-awake Local Anesthesia No Tourniquet (WALANT) Anesthesia in the Incidence of Complex Regional Pain Syndrome (CRPS) Following Common Hand Surgeries
Brief Title: Axillary Block or Wide-awake Local Anesthesia for Complex Regional Pain Syndrome (CRPS) Following Common Hand Surgeries
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Merve Dursun Savran, MD, MD, Principal Investigator, Ankara University
Other Study IDs: Axillary block vs Walant
Record Dates: First submitted 2025-03-01; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: CRPS; Walant; Axillary Block
Keywords: CRPS; flare reaction; WALANT; axillary block
MeSH Terms: interventions — Surgical Procedures, Operative; Anesthesia, Conduction; Anesthesia, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- WALANT: Patients operated under WALANT (wide awake local anesthesia without tourniquet)
  Interventions: Procedure: Surgery for Dupuytren contracture (DC), DeQuervain tenosynovitis (DQS), carpal tunnel syndrome (CTS), or trigger finger (TF); Procedure: Local Anesthesia
- RAAB: Patients operated under RAAB (regional anesthesia with axillary block)
  Interventions: Procedure: Surgery for Dupuytren contracture (DC), DeQuervain tenosynovitis (DQS), carpal tunnel syndrome (CTS), or trigger finger (TF); Procedure: Regional Anesthesia

INTERVENTIONS:
Procedure: Surgery for Dupuytren contracture (DC), DeQuervain tenosynovitis (DQS), carpal tunnel syndrome (CTS), or trigger finger (TF) — All of the patients were operated for Dupuytren contracture (DC), DeQuervain tenosynovitis (DQS), carpal tunnel syndrome (CTS), or trigger finger (TF). The study is two center study, one center has the routine of RAAB (regional anesthesia with axillary block) and the other has the routine of WALANT (wide awake local anesthesia no tourniquet) for the mentioned surgeries.
Procedure: Regional Anesthesia — Regional anesthesia with axillary block
  Groups: RAAB
Procedure: Local Anesthesia — Wide awake local anesthesia no tourniquet
  Groups: WALANT

SUMMARY:
Flare reaction, characterized by excessive erythema, stiffness, and edema postoperatively, can lead to complex regional pain syndrome (CRPS) when pain is present. This study compares flare and CRPS incidence following hand surgeries performed under regional anesthesia with axillary block (RAAB) and WALANT (Wide-Awake Local Anesthesia No Tourniquet).

DETAILED DESCRIPTION:
This two-center prospective study included patients undergoing Dupuytren contracture (DC), DeQuervain tenosynovitis (DQS), carpal tunnel syndrome (CTS), and trigger finger (TF) surgeries under RAAB or WALANT. Diagnostic criteria for flare and CRPS (pain, weakness, scar issues, erythema, and swelling) were assessed, and comorbidities were noted. The incidence of flare reactions and CRPS was compared for RAAB and WALANT.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with and operated on for Dupuytren contracture (DC),
* Patients diagnosed with and operated on for De Quervain tenosynovitis (DQS),
* Patients diagnosed with and operated on for carpal tunnel syndrome (CTS),
* Patients diagnosed with and operated on for trigger finger (TF)

Exclusion Criteria:

* Patients operated under general anesthesia,
* Patients operated with other types of regional anesthesia (eg: supraclavicular block),
* Patients operated with other types of local anesthesia (only prilocaine or bupivacaine)
* Patients less than 3 months follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: atients diagnosed with and operated on for Dupuytren contracture (DC), De Quervain tenosynovitis (DQS), carpal tunnel syndrome (CTS), or trigger finger (TF)
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
CRPS severity score (CSS) | Postoperative first month
  CRPS: Complex regional pain sydrome The CRPS Severity Score is a composite measure derived from multiple clinical findings, summed to provide a single score ranging from 0 to 16.
  The ccore is based on four major clinical domains, with each domain contributing 0 to 4 points, leading to a total possible score of 16 points.
  1. Sensory Symptoms (0-4 points) Allodynia (Pain due to a stimulus that does not normally provoke pain) Hyperalgesia (Increased pain response to a normally painful stimulus)
  2. Vasomotor Symptoms (0-4 points) Temperature asymmetry (≥1°C difference between affected and unaffected limb) Skin color changes (Mottled, red, cyanotic, or pale discoloration)
  3. Sudomotor / Edema Symptoms (0-4 points) Abnormal sweating (Hyperhidrosis or hypohidrosis) Edema (Swelling) in the affected area
  4. Motor / Trophic Symptoms (0-4 points) Motor dysfunction (Weakness, dystonia, tremors) Trophic changes (Altered nail growth, skin texture changes, or abnormal hair growth)
CRPS severity score (CSS) | Postoperative third month
  CRPS: Complex regional pain sydrome The CRPS Severity Score is a composite measure derived from multiple clinical findings, summed to provide a single score ranging from 0 to 16.
  The ccore is based on four major clinical domains, with each domain contributing 0 to 4 points, leading to a total possible score of 16 points.
  1. Sensory Symptoms (0-4 points) Allodynia (Pain due to a stimulus that does not normally provoke pain) Hyperalgesia (Increased pain response to a normally painful stimulus)
  2. Vasomotor Symptoms (0-4 points) Temperature asymmetry (≥1°C difference between affected and unaffected limb) Skin color changes (Mottled, red, cyanotic, or pale discoloration)
  3. Sudomotor / Edema Symptoms (0-4 points) Abnormal sweating (Hyperhidrosis or hypohidrosis) Edema (Swelling) in the affected area
  4. Motor / Trophic Symptoms (0-4 points) Motor dysfunction (Weakness, dystonia, tremors) Trophic changes (Altered nail growth, skin texture changes, or abnormal hair growth)

SECONDARY OUTCOMES:
Flare reaction | Postoperative first month
  Presence of Flare reaction. Evaluation based on Evans' criteria 0 - no reaction
  1. redness, stiffness, edema at the operation site
  2. symptoms beyond operation site
Flare reaction | Postoperative third month
  Presence of Flare reaction. Evaluation based on Evans' criteria 0 - no reaction
  1. redness, stiffness, edema at the operation site
  2. symptoms beyond operation site

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical Faculty, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Some individual personal data are pictures with identifiable elements of the patient.